CLINICAL TRIAL: NCT06705244
Title: Trans-nasal Sphenopalatine Ganglion Block Versus Ultrasound-guided Bilateral Greater and Lesser Occipital Nerve Block for Management of Post-Dural Puncture Headache After Spinal Anesthesia in Patients Undergoing Lower Abdominal Surgeries
Brief Title: Trans-nasal Sphenopalatine Ganglion Block Versus Ultrasound-guided Bilateral Greater and Lesser Occipital Nerve Block for Management of Post-Dural Puncture Headache.
Acronym: TNSPGB /GALONB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU MS141/2024
Record Dates: First submitted 2024-09-10; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-02

CONDITIONS: Post-Dural Puncture Headache
Keywords: Post dural Puncture headache; Trans-nasal Sphenopalatine Ganglion Block; Greater Occipital Nerve block; Lesser Occipital Nerve block; Spinal Anesthesia; Pain management; Ultrasound guided nerve blocks
MeSH Terms: conditions — Post-Dural Puncture Headache; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- trans-nasal sphenopalatine ganglion block (TNSGB) (Active Comparator)
  Interventions: Procedure: Trans-nasal sphenopalatine nerve block
- greater and lesser occipital nerve block (GALONB) (Active Comparator)
  Interventions: Procedure: Greater and lesser occipital nerve block

INTERVENTIONS:
Procedure: Trans-nasal sphenopalatine nerve block — The patient was placed supine with shoulders slightly elevated to flex the neck and extend the head.
  Then anterior nares were inspected for polyps, tumors, or significant septal deviation.
  Long cotton-tipped applicators saturated with lidocaine 2% were inserted into each naris, until properly seated in the posterior nasopharynx.
  These were left in place for 10 minutes to lubricate and anesthetize the mucous membrane, making the procedure more comfortable.
  Then a mixture of 3 mL of 2 mL lidocaine 2% plus 1 mL dexamethasone 4 mg were injected through the applicators in the sphenopalatine area in each nostril.
  Then the patient was positioned sitting and pain assessments were recorded.
  Arms: trans-nasal sphenopalatine ganglion block (TNSGB)
Procedure: Greater and lesser occipital nerve block — The back of the head was sterilized with an antiseptic solution and the landmarks at the base of the skull were identified while the patient in the prone position.
  The landmarks were located on the medial third of a line drawn from occipital protuberance to mastoid process. At this level, the greater and lesser occipital nerves lie along the superior nuchal line medial to the occipital artery, halfway between the occipital protuberance and mastoid process.
  Under Ultrasound guidance, the skin was infiltrated with 1-2 mL of lidocaine 2%, using a 25-gauge needle. Then the block was performed in this area with a mixture of 3 mL of 2 mL lidocaine 2% plus 1 mL dexamethasone 4 mg to block greater and lesser occipital nerves. Then the procedure was repeated on the other side.
  After the procedure, the presence of bilateral occipital numbness was confirmed after 30 minutes. The patient was then positioned sitting and pain scoring was assessed.
  Arms: greater and lesser occipital nerve block (GALONB)

SUMMARY:
Post-Dural Puncture Headache (PDPH) is a complication associated with spinal anesthesia. While conventional treatments are available, the Epidural Blood Patch (EBP) is considered the gold standard. Other less invasive interventions, such as Sphenopalatine Ganglion (SPG) block and Greater Occipital Nerve (GON) block, have also been used to treat PDPH. The trans-nasal approach is a non-invasive, low-risk technique that can be performed at the bedside without imaging tools.

The Lesser Occipital Nerve Block (LONB) is often used in conjunction with the GONB to address headaches in the lateral occipital region.

This study aims to compare the efficacy of trans-nasal sphenopalatine ganglion block (TNSGB) versus Greater and Lesser Occipital Nerve Block (GALONB) guided by ultrasound in relieving PDPH and its symptoms, as well as to assess patient satisfaction with the interventions.

Conducted at Ain Shams University Hospitals with approval from the medical ethical committee, the study included 50 participants (25 per group) who were ASA class I or II candidates for spinal anesthesia undergoing elective lower abdominal surgeries. Participants were randomly assigned to two groups:

* Group TNSGB: Received a trans-nasal sphenopalatine ganglion block using cotton-tipped applicators inserted trans-nasally until positioned in the posterior nasopharynx.
* Group GALONB: Received a Greater and Lesser Occipital Nerve Block under ultrasound guidance to identify nerves, foramina, vascular structures, and their course.

Patient satisfaction was evaluated using a 5-point Likert scale. The analgesic efficacy of TNSGB versus GALONB was assessed using a Numeric Rating Scale (NRS) at 0, 30 minutes, 1, 2, 3, 6, 12, 24, and 48 hours after treatment.

Adverse events, the need for rescue analgesia, and other therapeutic interventions were also recorded.

DETAILED DESCRIPTION:
* Type of Study:

Exploratory single-blind randomized comparative trial. (Only the data collection personnel were blinded to the group assignment).

• Study Settings: Ain Shams University Hospitals.

* Study Period:

  6 months
* Study Population:

All patients included in this study met the International Headache Society criteria for diagnosis of PDPH, as follows:

1. headache that:

   a) worsens within 15 minutes of sitting or standing; b) improves within 15 minutes after lying down; c) must have one of the following associated manifestations of: neck stiffness, tinnitus, hypoacusis, or photophobia;
2. dural puncture has been performed;
3. headache develops within 5 days after dural puncture.

   The headache should have persisted for at least two days and must have been intractable to conservative treatment with fluids, caffeine, paracetamol, and other nonopioid analgesics.

   Failure of conservative management was defined as headache score > 4/10 on a numerical rating scale (NRS) when the patient assumed an upright position.

   -Inclusion Criteria: Physical status: ASA 1 or 2 and candidates for spinal anesthesia undergoing elective lower abdominal surgeries.

   Age group: 18-45 years. Sex: Both sexes Body mass index of less than 35 kg/m2 -Exclusion Criteria: Declining to give written informed consent. History of allergy to the medications used in the study. Contraindications to regional anesthesia (including coagulopathy, and local infection).

   Psychiatric disorder and/or Drug Addiction. American Society of Anesthesiologists (ASA) Physical Status Class III and more. Moderate to severe hepatic and renal diseases. Emergency surgeries. Nasal septal deviation, Nasal deformity and/or nasal bleeding. Had received opioids less than 12 hours before study inclusion. History of migraines or persistent headaches.

   •Sampling Method: Patients fulfilling inclusion criteria will be randomly divided into two groups using their computer-generated random numbers.

   •Sampling Size: An exploratory study will be conducted that includes at least 50 participants (25/group) to compare the efficacy of trans-nasal sphenopalatine ganglion block (TNSGB) and greater and lesser occipital nerve block (GALONB) to relieve PDPH and its associated symptoms.

   •Ethical Considerations: The study will be performed after ethical committee approval and informed consent from the patients after full explanation of the procedure, possible side effects and complications.

   Informed written consent was taken from all patients after explaining the study procedure in detail.

   • Study Procedure:

   - Pre-operative Settings: All patients will have the same preoperative preparation and anesthetic technique. History and general examination will be done to all patients and routine investigations will be done preoperatively as laboratory investigations (complete blood picture, bleeding time, INR, partial thromboplastin-time, and blood chemistry as liver and kidney function tests). Age, weight, and sex will be recorded.

   - Intra-operative Settings: Inside the operating room/ward, intravenous access will be inserted, monitor connected and baseline non-invasive blood pressure (NBP), heart rate (HR), electrocardiography (ECG) and oxygen saturation (SpO2) will be measured.

   Patients were randomly allocated into 2 groups.

   o TNSPGB Group: The patient was placed supine with shoulders slightly elevated to flex the neck and extend the head.

   Then anterior nares were inspected for polyps, tumors, or significant septal deviation.

   Long cotton-tipped applicators saturated with lidocaine 2% were inserted into each naris, until properly seated in the posterior nasopharynx.

   These were left in place for 10 minutes to lubricate and anesthetize the mucous membrane, making the procedure more comfortable.

   Then a mixture of 3 mL of 2 mL lidocaine 2% plus 1 mL dexamethasone 4 mg were injected through the applicators in the sphenopalatine area in each nostril. (Youssef et al., 2021) Then the patient was positioned sitting and pain assessments were recorded. o GALONB Group: The back of the head was sterilized with an antiseptic solution and the landmarks at the base of the skull were identified while the patient in the prone position.

   The landmarks were located on the medial third of a line drawn from occipital protuberance to mastoid process. At this level, the greater and lesser occipital nerves lie along the superior nuchal line medial to the occipital artery, halfway between the occipital protuberance and mastoid process.

   Under Ultrasound guidance, the skin was infiltrated with 1-2 mL of lidocaine 2%, using a 25-gauge needle. Then the block was performed in this area with a mixture of 3 mL of 2 mL lidocaine 2% plus 1 mL dexamethasone 4 mg to block greater and lesser occipital nerves. Then the procedure was repeated on the other side.

   After the procedure, the presence of bilateral occipital numbness was confirmed after 30 minutes. The patient was then positioned sitting and pain scoring was assessed.

   *Both blocks will be done and/or supervised by an expert all through.

ELIGIBILITY:
Inclusion Criteria:

Physical status: ASA 1 or 2 and candidates for spinal anesthesia undergoing elective lower abdominal surgeries.

Age group: 18-45 years. Sex: Both sexes Body mass index of less than 35 kg/m2

Exclusion Criteria:

Declining to give written informed consent. History of allergy to the medications used in the study. Contraindications to regional anesthesia (including coagulopathy, and local infection).

Psychiatric disorder and/or Drug Addiction. American Society of Anesthesiologists (ASA) Physical Status Class III and more. Moderate to severe hepatic and renal diseases. Emergency surgeries. Nasal septal deviation, Nasal deformity and/or nasal bleeding. Had received opioids less than 12 hours before study inclusion. History of migraines or persistent headaches.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | After 48 hours
  Patients were asked to evaluate their satisfaction regarding the received intervention through 5-point Likert scale (1 = very satisfied, 2 = satisfied, 3 = neither satisfied nor dissatisfied, 4 = dissatisfied, 5= very dissatisfied).

SECONDARY OUTCOMES:
the analgesic efficacy of the TNSPGB versus GALONB for treatment of PDPH | at baseline 0, at 30 minutes, 1 hour , 2 hours, 3 hours, 6 hours, 12 hours, 24hours and 48 hours after treatment.
  using a Numeric Rating Scale (NRS) from 0 to 10
Need for rescue analgesia | after 4 hours of given intervention
  Need for rescue analgesia If pain score on Numeric rating scale = or > 4

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uyar Turkyilmaz E, Camgoz Eryilmaz N, Aydin Guzey N, Moraloglu O. Bilateral greater occipital nerve block for treatment of post-dural puncture headache after caesarean operations. Braz J Anesthesiol. 2016 Sep-Oct;66(5):445-50. doi: 10.1016/j.bjane.2015.03.004. Epub 2016 Jan 21. PMID 27591456
- [Background] Goncalves LM, Godinho PM, Duran FJ, Valente EC. Sphenopalatine ganglion block by transnasal approach in post-dural puncture headache. J Clin Anesth. 2018 Aug;48:50. doi: 10.1016/j.jclinane.2018.05.006. Epub 2018 May 8. No abstract available. PMID 29751211
- [Background] Nair AS, Kodisharapu PK, Anne P, Saifuddin MS, Asiel C, Rayani BK. Efficacy of bilateral greater occipital nerve block in postdural puncture headache: a narrative review. Korean J Pain. 2018 Apr;31(2):80-86. doi: 10.3344/kjp.2018.31.2.80. Epub 2018 Apr 2. PMID 29686805
- [Background] Youssef HA, Abdel-Ghaffar HS, Mostafa MF, Abbas YH, Mahmoud AO, Herdan RA. Sphenopalatine Ganglion versus Greater Occipital Nerve Blocks in Treating Post-Dural Puncture Headache after Spinal Anesthesia for Cesarean Section: A Randomized Clinical Trial. Pain Physician. 2021 Jul;24(4):E443-E451. PMID 34213869